CLINICAL TRIAL: NCT05926791
Title: Evaluation of the Photoprotective Effects of a SPF50+ Sunscreen on Photo-induced Cell Damage in Epidermal and Urine Samples, Following a Repeated Chronic Outdoor Sun Exposure in Healthy Adults
Brief Title: Photoprotective Effects of a SPF50+ Sunscreen on Skin Genotoxicity Induced by Repeated Chronic Outdoor Sun Exposure
Status: Completed | Type: Observational
Sponsor: Pierre Fabre Dermo Cosmetique (Industry)
Responsible Party: Sponsor
Other Study IDs: DNAOUTDOOR
Record Dates: First submitted 2023-01-12; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Sun Damaged Skin
Keywords: Sunscreen; Chromametry and pigmentation; Suction blister; Liquid chromatography-High resolution Mass spectrometry; Mass spectrometry lipid analysis; Urine
MeSH Terms: interventions — Cosmetics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Educated group with product: Subjects receiving the SPF50+ sunscreen product and a targeted educational action
  * Route of administration: Topical
  * Application duration: from 5 up to 21 days
  * Application modalities: The investigational product will be applied during the outdoor sun exposure on all exposed parts of the body (face and body). The investigational product will be applied in sufficient amount to cover the exposed areas (2mg/cm2 recommended), 15 to 30 minutes before each sun exposure. The product should be reapplied as many times as required during sun exposure (systematic reapplication of the product after sweating and/or swimming and/or wiping).
  Interventions: Other: Cosmetic product
- Control group: Subjects receiving neither product nor targeted education

INTERVENTIONS:
Other: Cosmetic product — The educated group receives the cosmetic product SPF50+ according to the randomization list established at V1 and returns the products at V2
  Groups: Educated group with product

SUMMARY:
Between 2 and 3 million non-melanoma skin cancers and 132,000 melanoma skin cancers occur globally each year. Sun protection continues to be a major public health issue and has always been a priority research area for Pierre Fabre laboratories. The involvement of ultraviolet radiation of the solar spectrum in skin carcinogenesis is well known, through its ability to damage the DNA of skin cells and the induction of oxidative processes.

The aim of this exploratory study is to perform the quantification of:

* DNA photoproducts excised from the genome by the biological repair systems in urine samples
* cellular DNA damage in the epidermis following chronic exposure to natural sunlight.

This study will allow us to better understand and quantify the benefit of sunscreens on photoinduced cellular damage and their elimination in urine.

DETAILED DESCRIPTION:
This trial is a monocentric, exploratory, randomized, controlled, open-label, parallel-group study conducted in healthy adult subjects.

The target population consists of subjects who are accustomed to using few products or using low protection index during sun exposure.

The study area is the whole body for sun exposure. The target areas are the face and forearms for the samplings and measurements.

In this design, in order not to impose any strong constraint to the subjects in terms of sun exposure, the duration of the exposure period is left free and can vary between 5 and 21 days. Within this window, subjects can freely determine their sun exposure episodes (choice of time slot, number and duration). However, subjects have to expose themselves for at least 3 hours /day, for 5 days in the week prior to visit 2 (which will be scheduled no more than 3 days after their last sun exposure).

The study includes 3 visits:

* Visit 1: Inclusion (D1)
* Visit 2: Intermediate visit (D7 to D39)
* Visit 3: Wound healing evaluation and end of study (V2 + 15 days +/- 2 days)

The period of outdoor sun exposure varies between 5 and 21 days depending on the duration planned by the subjects themselves. This is also the duration of application of the investigational product for the subjects in group 1.

Visit 1 can be performed up to 15 days before the beginning of the sun exposure period and visit 2 up to 3 days after the last sun exposure.

The duration of participation for a subject varies between 20 and 56 days (from inclusion to the end of the study).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged between 18 and 55 years included
* Subject with a habit of using little or no sunscreen products with low protection index (SPF < 25) during sun exposure.
* Subject's commitment to have a self-reported sun exposure of at least 3 hours per day for the 5 days of their last week of vacation
* Subjects agreeing not to expose themselves to UVs (natural or artificial) before the planned outdoor sun exposure period

Exclusion Criteria:

1. - Criteria related to the population:

   * Smoker of more than 10 cigarettes per day containing nicotine, paper and/or electronic cigarette equivalent
   * Subject having received on study areas artificial UV exposure or excessive, prolonged, and unprotected exposure to natural sunlight within the 4 weeks before the inclusion visit or planning one during the study
   * Subject having performed excessive and prolonged physical activity (e.g. trail, long distance running, race…) within 7 days before the inclusion visit
2. - Criteria related to the diseases / skin condition:

   * Subject with a known history of photosensitivity (toxic, allergic)
   * Subject with a known personal or family history of skin cancer
   * Subject having hereditary or acquired disorders of hemostasis.
3. - Criteria related to the treatments and/or products:

   * Physical treatment (radiotherapy, phototherapy, chemical peeling, laser, ...) on the study area within 4 weeks before the inclusion visit or planned during the study.
   * Systemic or topical treatment applied on the study area (e.g. anti-allergic, anti-inflammatory treatment) within two weeks before the inclusion visit, ongoing or planned during the study and likely to interfere with the study according to the investigator's assessment
   * Use of anti-aging products (containing retinoids and / or α-hydroxy acids) on the target areas (face and/or forearms) in the 2 weeks before the inclusion visit.
   * Systemic or topical treatment with photosensitizing or phototoxic potential (NSAIDs, antihistamines, psychotropic drugs, antidepressants, anti-migraine drugs, cyclines, quinolone, antibiotics, beta-blockers, etc.), taken or applied to the study area within the previous weeks, ongoing or planned during the study, and likely to interfere with the study according to the investigator's assessment
   * Subject taking creatine dietary supplements and/or practicing prolonged fasting

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects will be recruited from the investigation centre's panel. The participants will be selected on the basis of inclusion and non-inclusion criteria specific to the study and on their ability to comply with the constraints required by the protocol. The participants will be definitely included in the study after a specific interview and a clinical examination
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Change in photoinduced DNA damage products in urine samples before and after outdoor sun exposure | Change from baseline (day 1) to visit 2 (occuring between day 7 to 39 depending on the duration of sun exposure)
  Quantitative analysis of photoinduced DNA damage products by high performance liquid chromatography-coupled to tandem Mass Spectrometry (HPLC/MS-MS)
Number of CPD (Cyclobutane Pyrimidine Dimer) lesions in epidermal samples collected from the forearm following the outdoor sun exposure period | Day 7 to 39 (depending on the duration of sun exposure)
  Number of CPD (Cyclobutane Pyrimidine Dimer) lesions in epidermal samples by high performance liquid chromatography-coupled to tandem Mass Spectrometry (HPLC/MS-MS)
Change in colorimetric parameters before and after outdoor sun exposure | Change from baseline (day 1) to visit 2 (between day 7 to 39 depending on the duration of sun exposure)
  Colorimetric parameters assessed by chromametry on the face and forearm
Change in pigmentation parameters before and after outdoor sun exposure | Change from baseline (day 1) to visit 2 (between day 7 to 39 depending on the duration of sun exposure)
  Pigmentation parameters assessed by Multispectral analysis on the face and forearms
Change in cellular damages before and after outdoor sun exposure | Change from baseline (day 1) to visit 2 (between day 7 to 39 depending on the duration of sun exposure) up to visit 3 ( between day 20 to 56)
  Cellular damage assessed by Mass spectrometry lipid analysis in D-Squame samples collected on the face and forearm before and after outdoor sun exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Research Center, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided